CLINICAL TRIAL: NCT06119698
Title: Randomized, Hybrid Type 1 Effectiveness-implementation Trial of GetActive+ vs Treatment as Usual; iHOPE Study
Brief Title: Improving Health for Older Adults With Pain Through Engagement
Acronym: iHOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P000782
Record Dates: First submitted 2023-10-17; First posted 2023-11-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Musculoskeletal Pain
Keywords: Older adults; Mind-body intervention; Chronic pain; ActiGraph; Community health center; Physical function
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GetActive+ (Experimental): A mind-body program focused on increasing physical and emotional function in older adults with chronic musculoskeletal pain
  Interventions: Behavioral: GetActive+
- Treatment as usual (No Intervention): Treatment as Usual (TAU) includes traditional primary care management of chronic pain.

INTERVENTIONS:
Behavioral: GetActive+ — This is a 10-week group mind body program focused on improving self-reported physical activity, performance-based physical activity, and ambulatory step count by combining mind body skills tailored for individuals with chronic pain, with gradual increase in walking using quota based pacing and goal setting, adapted specifically for older adults from a medically underserved location.
  Arms: GetActive+

SUMMARY:
The goal of this project is to conduct a randomized, hybrid type 1 effectiveness-implementation trial (N=200) to evaluate the effectiveness and implementation of a 10-week mind-body and walking program (GetActive+) vs treatment as usual (TAU). The investigators will test for improvements in self-reported, performance-based (i.e., six-minute walk test), and objective (i.e., step-count) physical function, emotional function, as well as feasibility, acceptability and implementation markers. Participants will complete measures at baseline (0 weeks), post-intervention (1 week after intervention completion), and 6-month follow-up.

This study will receive support from and inclusion in the HEAL Initiative (https://heal.nih.gov/).

DETAILED DESCRIPTION:
The aim of this phase is to conduct a randomized, hybrid type 1 effectiveness-implementation trial (N=200) to evaluate the effectiveness and implementation of GetActive+ vs TAU on the following outcomes.

Aim 1: Self-reported physical function at 10 weeks (primary). Aim 2: Self-reported physical function at 6 months, performance based (6-minute walk test), and objective (step-count) physical function, as well as self-reported emotional function, pain, social support and loneliness at 10 weeks and 6 months.

Aim 3: Feasibility, acceptability, fidelity and adoption at patient, provider, and organization levels based on Proctor's implementation framework.

The investigators will enroll N=200 older adults with chronic pain from Revere HealthCare Center and MGH Broadway Primary Care in Revere. The GetActive+ program used in the Randomized Controlled Trial (RCT) will incorporate mind-body skills, cognitive behavioral and physical restoration skills (e.g., quota-based pacing) to help individuals increase self-reported, performance based and objective (step count) physical function. This program will teach participants four core skills: 1) weekly goal setting for gradual increase in time spent walking paired with activities of daily living that are meaningful and important to participants (i.e. walk instead of drive to the store; walk to the park with kids); 2) quota-based pacing (increasing walking goal gradually non-contingent of pain); 3) mind-body skills (e.g., diaphragmatic breathing to manage intense pain flares and pain anxiety; progressive muscle relaxation to increase body awareness and reduce reactivity to pain sensations; mindfulness exercises to understand the transience of pain and change one's relationship with it; self-compassion when falling short of set goals); and 4) understand the downward spiral (e.g. how reducing activity perpetuates pain and disability), correct myths about pain or unhelpful pain-related thoughts that interfere with meeting program goals. Participants will be encouraged to complete their homework (logs for mind-body practice, physical activities) each day. Participants will be given the option to receive homework and session reminders via text messages from study staff. This between-session contact will focus on increasing treatment adherence, maintaining engagement, and session reminders. The investigators will run groups primarily in English with additional groups in Spanish.

Baseline assessments, post-intervention assessments and 6-month follow up assessments will include the 6MWT, objective step count via ActiGraph, and self-reported measures including physical function, emotional function, pain, social support, and loneliness while accounting for clinical, demographic, and social determinants of health.

ELIGIBILITY:
Inclusion Criteria:

1. Older Adults (i.e., age >=55)
2. Diagnosed musculoskeletal chronic pain of any type (e.g., pain > 3 months)
3. Pain score >=4 (moderate) on the Numerical Rating Scale
4. Cognitively able to participate as measured by the Short Portable Mental Health questionnaires (e.g., <4 errors)
5. Self-reported ability to complete the 6-minute walk test including with assistive devices
6. Patient at Revere HealthCare Center or MGH Broadway Primary Care in Revere who is cleared for participation by medical staff
7. English or Spanish fluency and literacy

Exclusion Criteria:

1. Current serious medical illness that is expected to worsen in the next 6 months (e.g., cancer)
2. Individuals who are unwilling or unable to comply with study procedures including wearing a smartwatch
3. Active suicidal ideation with plan or intent
4. Active and untreated serious mental health or substance use disorder

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Physical function - self-report | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total) - Measure time point of 10 weeks is considered for primary outcome.
  Patient-Reported Outcomes Measurement Information System (PROMIS) v2.0 Physical Functioning Short Form 6b; assesses ability to carry out activities that require physical actions, ranging from self-care to work. Scores range from 6 to 30, with higher scores indicating greater physical function.

SECONDARY OUTCOMES:
Physical function - objective | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Average step count with wrist-worn ActiGraph wGT3X-BT; collects average step count for 4-7 days.
Physical function - performance-based | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  6-minute walk test (6MWT); measures the total distance in meters covered by an individual in 6 minutes, with greater distances covered indicating better physical function.
Pain Intensity and Severity | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Brief Pain Inventory - Short Form (BPI-SF); assesses pain severity and interference. Scores range from 0 to 10, with higher scores indicating more severe pain severity or interference.
Pain Intensity and Interference | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Pain, Enjoyment of Life and General Activity (PEG) Scale; measures pain intensity and pain interference in the enjoyment of life and activities of daily living. Scores range from 0 to 10, with higher scores indicating more severe pain and related interference.
Depression | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Patient Health Questionnaire - 8 (PHQ-8); assesses depressive symptoms. Scores range from 0 to 24, with higher scores indicating more severe depressive symptoms.
Anxiety | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Generalized Anxiety Disorder - 7 (GAD-7); measures anxiety symptoms. Scores range from 0 to 21, with higher scores indicating greater anxiety.
Impression of Change | Post-Intervention
  Patient Global Impression of Change (PGIC); assesses subjective changes in response to the intervention. Scores range from 0 to 6, with higher scores indicating worse outcomes.

OTHER OUTCOMES:
Quota-based Pacing | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  4-item subsection of the Activity Pacing Questionnaire; measures ability to pace. Scores range from 4 to 20, with higher scores indicating increased quota-based pacing.
Pain Catastrophizing | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Pain Catastrophizing Scale (PCS); assesses magnification, helplessness, and rumination associated with the ability to cope with pain. Scores range from 0 to 52, with higher scores indicating increased pain catastrophizing.
Mindfulness | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Applied Mindfulness Process Scale (AMPS); assesses mindfulness use in daily life. Scores range from 0 to 60, with higher scores indicating greater utilization of mindfulness.
Current Status | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Measure of Current Status (MOCS); assesses healthy coping skills. Scores range from 0 to 52, with higher scores reflecting a stronger ability to recognize and cope with stress.
Self-Compassion | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Self-Compassion Scale - Short Form (SCS-SF); assesses the ability to practice self-compassion. Scores range from 1 to 5, with higher scores associated with lower levels of self-compassion.
Social Support | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Interpersonal Support Evaluation List - 12 (ISEL-12); measures perceptions of social support. Scores range from 12 to 48, with higher scores indicating stronger social support.
Loneliness | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  University of California Los Angeles - 3 Loneliness Scale (UCLA-3); measures loneliness in relational connectedness, social connectedness, and social isolation. Scores range from 3 to 9, with higher scores indicating greater social isolation.
Fear of Pain | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Tampa Scale for Kinesiophobia - 11 (TSK-11); assesses fear of pain and activities that cause pain. Scores range from 11 to 44, with higher scores reflecting more severe kinesiophobia.
Self-Efficacy for Exercise | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Self-Efficacy for Exercise (SEE); assesses an individual's beliefs in their ability to exercise three times per week for 20 minutes. Scores range from 0 to 90, with higher scores indicating higher confidence in exercising despite barriers.
Post Traumatic Stress Disorder | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Abbreviated Post-Traumatic Checklist-Civilian Version (PCL-C-6); assess current Post Traumatic Stress Disorder (PTSD) symptoms. Scores range from 6 to 30, with higher scores being suggestive of greater difficulties with post-traumatic stress.
Discrimination | Baseline
  Everyday Discrimination Scale - Short Version (EDS-S); assesses experiences of daily discrimination against minority populations. Scores range from 0 to 25, with higher scores indicating greater frequency of discriminatory experiences.
Stress | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Perceived Stress Scale - 4 (PSS-4); assesses stress perception levels. Scores range from 0 to 16, with higher scores indicating more severe stress.
Substance Use | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  Tobacco, Alcohol, Prescription medications, and other Substance use (TAPS); assess substance use behaviors. Each substance is scored individually from 0 to 4, with lower scores indicating more problematic substance use behaviors.
Sleep Duration | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  1-item of the Pittsburgh Sleep Quality Index (PSQI); assesses average sleep duration per night in the past month.
Sleep Disturbance | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  PROMIS v1.0 Sleep Disturbance - Short Form 6a; assesses duration and quality of sleep. Scores range from 6 to 30, with greater scores indicating higher sleep quality and more sleep disturbance.
Quality of Life Assessment | Baseline, Post-Intervention, 6-Month Follow Up (~9 months total)
  World Health Organization Quality of Life - 2 (WHOQOL-2); assesses satisfaction with health and quality of life. Scores range from 2 to 10, with higher scores indicating greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital; Christine Ritchie, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data file (e.g., blinded Excel with raw scores at each time point) Data dictionary Detailed protocol Analysis plan
Supporting Information: Study Protocol, SAP
Time Frame: Information is anticipated to be available 6 months after completion of the study.
Access Criteria: Data can be accessed in the Vivli data repository; no specialized tools will be need to view the data other than what is noted on the Vivli website. See above for details on what will be available to access.
URL: https://www.vivli.org

REFERENCES:
- [Background] Greenberg J, Lin A, Popok PJ, Kulich RJ, Edwards RR, Vranceanu AM. Getting Active Mindfully: Rationale and Case Illustration of a Group Mind-body and Activity Program for Chronic Pain. J Clin Psychol Med Settings. 2021 Dec;28(4):706-719. doi: 10.1007/s10880-020-09758-w. Epub 2021 Jan 19. PMID 33469845
- [Background] Grunberg VA, Greenberg J, Mace RA, Bakhshaie J, Choi KW, Vranceanu AM. Fitbit Activity, Quota-Based Pacing, and Physical and Emotional Functioning Among Adults With Chronic Pain. J Pain. 2022 Nov;23(11):1933-1944. doi: 10.1016/j.jpain.2022.07.003. Epub 2022 Jul 29. PMID 35914640
- [Background] Popok PJ, Greenberg J, Gates MV, Vranceanu AM. A qualitative investigation of activity measurement and change following a mind-body activity program for chronic pain. Complement Ther Clin Pract. 2021 Aug;44:101410. doi: 10.1016/j.ctcp.2021.101410. Epub 2021 May 2. PMID 33971485
- [Derived] Vonderheide C, Kilduff C, McDermott KA, Greenberg J, La Camera DE, Giraldo-Santiago N, Kurkul A, Alvarez-Frank N, Kim Y, Pasinski R, Gholston M; iHOPE Study Team; Ritchie CS, Vranceanu AM. Protocol for a hybrid type 1 effectiveness-implementation trial of a mind-body activity program for older adults with chronic pain in a medically underserved area: The iHOPE study. Contemp Clin Trials. 2025 Dec;159:108116. doi: 10.1016/j.cct.2025.108116. Epub 2025 Oct 24. PMID 41326265